CLINICAL TRIAL: NCT03310528
Title: Gastric Ultrasound for Estimation of the Aspiration Risk in High Aspiration-risk Surgical Patient Populations
Brief Title: Gastric Ultrasound for Estimation of the Aspiration Risk Study
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201602234; OCR18887 (Other: University of Florida)
Record Dates: First submitted 2017-10-04; First posted 2017-10-16 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Aspiration of Gastric Contents
Keywords: Aspiration risk; GI Endoscopy; Fasting guidelines; Delayed gastric emptying
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents; Gastroparesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obeyed fasting guidelines: Scheduled GI endoscopy procedure with planned oral-gastric tube placed. Complete interview questionnaire. Gastric ultrasound exam prior to upper GI endoscopy procedure.
  Interventions: Behavioral: Interview questionnaire; Procedure: Gastric ultrasound exam
- Did not obey fasting guidelines: Scheduled GI endoscopy procedure with planned oral-gastric tube placed. Complete interview questionnaire. Gastric ultrasound exam prior to upper GI endoscopy procedure.
  Interventions: Behavioral: Interview questionnaire; Procedure: Gastric ultrasound exam
- Trauma - obeyed fasting guidelines: Scheduled GI endoscopy procedure with planned oral-gastric tube placed. Complete interview questionnaire. Gastric ultrasound exam prior to upper GI endoscopy procedure.
  Interventions: Behavioral: Interview questionnaire; Procedure: Gastric ultrasound exam
- Trauma - did not obey fasting guidelines: Scheduled GI endoscopy procedure with planned oral-gastric tube placed. Complete interview questionnaire. Gastric ultrasound exam prior to upper GI endoscopy procedure.
  Interventions: Behavioral: Interview questionnaire; Procedure: Gastric ultrasound exam

INTERVENTIONS:
Behavioral: Interview questionnaire — Complete interview questionnaire regarding the composition and timing of their most recent food intake.
Procedure: Gastric ultrasound exam — Gastric ultrasound exam prior to upper GI endoscopy procedure.

SUMMARY:
The purpose of this research study is to look at the effectiveness of current anesthesia guidelines regarding food and drink prior to surgery in patients who are likely to have food and drink remain in their stomach longer than might ordinarily be expected.

DETAILED DESCRIPTION:
Examine the utility of ultrasound examination of the stomach in estimating aspiration risk in patient populations whose aspiration risk is currently poorly understood. Evaluate the applicability of current pre-surgical fasting guidelines in the same patient populations whose aspiration risk is poorly understood.

Evaluate the residual gastric contents in patients presenting for upper GI endoscopy procedures who have adhered to pre-operative fasting guidelines. Evaluate the residual gastric contents in patients presenting for upper GI endoscopy procedures who have not adhered to pre-operative fasting guidelines. Only patients expected to have an oral-gastric tube placed during upper GI endoscopy procedure will be included. Both groups will be evaluated to learn if their residual gastric contents conform to currently-accepted standards for low aspiration risk.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for upper GI endoscopy procedures or surgical repair of a trauma- related injury
* Expected to have an oral-gastric tube placed as part of scheduled procedure
* Willing to undergo an ultrasound exam
* Patients ≥ 18 years of age

Exclusion Criteria:

* Unwilling to undergo an ultrasound exam
* Oral-gastric tube placement is not indicated
* Oral-gastric tube placement is contraindicated
* Pregnant patients and patients from defined vulnerable populations (ex. pediatric patients, mentally handicapped patients, prisoners, etc.)
* Surgical trauma patients who are not expected to have an OG tube placed during surgery
* Patients with history of gastric bypass surgery
* Patients that are gastrostomy tube dependent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for upper GI endoscopy and/or endoscopic retrograde cholangiopancreatogram (ERCP), expected to have an oral-gastric tube placed as part of scheduled procedure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
Changes in gastric content volume between the four groups assessed by ultrasound examination | Up to 12 hours
  Evaluate the residual gastric contents in patients presenting for upper GI endoscopy procedures to learn if their residual gastric contents conform to currently-accepted standards for low aspiration risk.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Smith, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- United States, Florida UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No